CLINICAL TRIAL: NCT07281833
Title: An Interventional, Open-label, Phase III Study to Evaluate the Safety, Efficacy, and Impact on Quality of Life of Capivasertib Alongside Standard-of-care Endocrine Treatment in Patients With HR+/HER2- Advanced Breast Cancer and Progression on Prior Endocrine-based Treatment
Brief Title: Phase III Study to Evaluate the Safety, Efficacy, and Impact on Quality of Life of Capivasertib Alongside Standard-of-care Endocrine Treatment in Patients With HR+/HER2- Advanced Breast Cancer and Progression on Prior Endocrine-based Treatment
Acronym: CAPIcorn
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: West German Study Group (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WSG-AM14 (CAPIcorn)
Record Dates: First submitted 2025-11-19; First posted 2025-12-15 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer; HR-positive Breast Cancer; Advanced Breast Cancer; Metastatic Breast Cancer; HER2-negative Breast Cancer
Keywords: breast cancer; advanced, metastatic; metastatic; progression; HR+; HER2-; capivasertib; eHealth; ePRO
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis; Disease Progression | interventions — capivasertib

STUDY DESIGN:
Intervention Model Description: This is a multicentre, interventional, prospective, one-armed, open-label, phase-III-trial to evaluate the use of capivasertib in patients with HR+/HER2- advanced breast cancer and progression on prior endocrine-based treatment
  The study will consist of:
  A. a recruitment phase, 24 months, during which the patients are screened and enrolled B. a study treatment and follow-up phase of up to 60 months until end of study, dependent on timepoint of enrolment in the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Capivasertib (Experimental): 2x400 mg, peroral, for 4 days, followed by 3 days off treatment
  Interventions: Drug: Capivasertib

INTERVENTIONS:
Drug: Capivasertib — 2x400 mg, peroral, for 4 days, followed by 3 days off treatment

SUMMARY:
This is a multicentre phase-III-trial to evaluate the use of capivasertib in patients with HR+/HER2- advanced breast cancer and progression on prior endocrine-based treatment.

The goal of this study is

1. To evaluate benefit of capivasertib regarding time to next treatment (TTNT1) - i.e., time "on treatment" with capivasertib.
2. To evaluate the benefits of patient reported outcome(PRO)-adherence regarding the deterioration of quality of life (DQoL)-free interval.

There is no active comparison group but a historical control group consisting of data of patients treated within the CAPItello-291-study..

Participants will take capivasertib accompanied by standard of care endocrine treatment and are asked to document ther quality of life on standardised questionnaires. Optionally, patients can use eHealth support via their own smart phones.

DETAILED DESCRIPTION:
Trial type: Interventional Clinical indication: HR+/HER2- advanced breast cancer under progress

IMP: capivasertib (CAPI) AxMP: fulvestrant (FULV) AxMP: GnRH agonists (GnRH)

Dose and route of administration: IMP: 2x400 mg, peroral, for 4 days, followed by 3 days off treatment AxMP FULV: 500 mg, intramuscular, every 28 days AxMP GnRH-agonist: according to SmPC of the medicinal product used

Treatment arm 1

* capivasertib (CAPI)
* with and without eHealth support (CANKADO PRO-active)

Type of control:

* No active control or comparator for Arm 1-treatment
* Historical study data from CAPItello-291 study

Trial blinding: Not applicable; open-label Number of trial participants: N=250 patients (Screening of about 600 patients expected to recruit 250 patients with alterations of the PIK3CA/AKT1/PTEN biomarkers)

Estimated enrolment period: 24 months Estimated duration of trial: Recruitment interval (expected 24 months) plus minimum 36 months follow-up (after LPI).

* Expected FPI: Q4 / 2024 - Q1 / 2025
* EOS: Q1 / 2030 Duration of participation: All patients will be followed-up from time point of inclusion until global End of Study (EOS) or death, whatever happens first.

Length of study treatment per patient: Capivasertib (CAPI) will be started after inclusion in the study and be administered until next progression, death, until any unbearable medical or other reason occurs that requires end of study for the patient, or global End of Study (EOS), whatever happens first.

ELIGIBILITY:
Inclusion Criteria:

1. Females (≥18 years, pre-, peri- or post-menopausal) and males (≥18 years) at the time of signing the informed consent form

   a. Pre-menopausal (and peri-menopausal, i.e., those that do not meet the criteria for post menopausal defined below) women can be enrolled if amenable to treatment with an GNRH agonist. Patients are to have commenced concomitant treatment with GNRH agonist prior to or on Cycle 1, Day 1 and must be willing to continue it for the duration of the study.

   b. Post-menopausal women are defined as: i. aged ≥60 years of age, OR ii. aged <60 years of age and amenorrhoeic for at least 12 months following cessation of all exogenous hormonal treatments/chemotherapy/ovarian suppression/tamoxifen or similar. These patients should also have serum oestradiol and follicle stimulating hormone (FSH) levels confirmed as being within the standard laboratory reference range for post-menopausal females, OR iii. documented bilateral oophorectomy.
2. Histologically confirmed HR+/HER2- breast cancer determined from the most recent tumour sample (primary or metastatic) as per WHO classification. To fulfil the requirement of HR+ disease, a breast cancer must express ER with or without co-expression of progesterone receptor.

   Therefore, tumours must be:

   a. ER+ defined as ≥1% of tumour cells stain positive for ER on immunohistochemistry (IHC) or, if no percentage is available, then an Allred IHC score of ≥3/8, b. Progesterone receptor positive defined as ≥1% of tumour cells stain positive for progesterone receptor on IHC or, if no percentage is available, then an Allred IHC score of ≥3/8; or progesterone receptor negative defined as <1% of tumour cells stain positive for progesterone receptor on IHC or, if no percentage is available, then an Allred IHC score of ≤2/8; or progesterone receptor unknown, and c. HER2- defined as 0 or 1+ intensity on IHC, or 2+ intensity on IHC and no evidence of amplification on in situ hybridisation (ISH), or if IHC not done, no evidence of amplification on ISH.
3. Metastatic or locally advanced disease with radiological or objective evidence of recurrence or progression (the cancer should have shown progression during or after most recent therapy); locally advanced disease must not be amenable to resection with curative intent (patients who are considered suitable for surgical or ablative techniques following potential down-staging with study treatment are not eligible).
4. Patients are to have received treatment with an ET (endocrine-based therapy) containing regimen (single agent or in combination) and have:

   a. Radiological evidence of breast cancer recurrence or progression while on, or within 12 months of the end of (neo)adjuvant treatment with an ET, OR b. Radiological evidence of progression while on prior ET administered as a treatment line for locally advanced or metastatic breast cancer (this does not need to be the most recent therapy).
5. Presence of one or more of the PIK3CA/AKT1/PTEN biomarkers, preferably determined in tumour tissue*
6. Decision to newly initiate capivasertib
7. Informed consent provided by patient prior to participation in the trial and before initiation of any study-specific measures
8. A. Female patients of childbearing potential at inclusion must have a negative pregnancy test (serum) and additionally, - surgically sterile, - carry an intrauterine device (combined with a barrier method),

   * having received a bilateral tubal ligation/occlusion (combined with a barrier method),
   * or using a highly effective method of contraception for the duration of the study (from the time they sign consent) and for 3 months after the last dose of capivasertib / GNRH and for 2 years after the last dose of fulvestrant to prevent pregnancy.
   * Total/true abstinence When the patient refrains from any form of sexual intercourse and this is in line with their usual and/or preferred lifestyle; this must continue for the duration of the study and for 3 months after the last dose of capivasertib/ GNRH and for 2 years after the last dose of fulvestrant to prevent pregnancy.
   * Vasectomised sexual partner (with participant assurance that partner received post-vasectomy confirmation of azoospermia) combined with a barrier method or sexual partner with bilateral orchiectomy
   * Hormonal contraception is not acceptable.

8. B. Male patients must either be

* surgically sterile
* or using an highly effective method of contraception for the duration of the study (from the time they sign consent) and for 4 months after the last dose of capivasertib/ GNRH and for 2 years after the last dose of fulvestrant to prevent pregnancy in a partner.
* Sexually abstinent men (i.e., refraining from heterosexual intercourse during the entire study duration) must continue for 4 months after the last dose of capivasertib/ GNRH and for 2 years after the last dose of fulvestrant to prevent pregnancy in a partner.
* Male patients who intend to be sexually active with a woman of childbearing potential, must use a condom plus spermicide upon entering the study and until 4 months after the last dose of capivasertib and for 2 years after the last dose of fulvestrant to prevent pregnancy in a partner.
* Highly effective methods of contraception should be considered in female partners of men taking capivasertib plus fulvestrant who are of childbearing potential.

  9. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 with no deterioration over the previous 2 weeks and life expectancy of ≥12 weeks

  *A list of eligible alterations and test procedures is provided in the protocol.

Exclusion Criteria:

* Patients eligible for inclusion in this study must not meet any of the following criteria:

  1. Absence of an alteration in the PIK3CA/AKT1/PTEN biomarkers
  2. Previous enrolment in the present study
  3. Participation in another clinical study with any investigational medicinal product and still on IMP treatment or have participated in an interventional study that remains blinded
  4. A disease burden that makes the patient ineligible for endocrine-based therapy per the investigator's best judgement (e.g., symptomatic visceral disease that is potentially life threatening in the short-term)
  5. Known history of drug or alcohol abuse within 1 year of screening
  6. Except for alopecia, any unresolved toxicities from prior therapy CTCAE Grade ≥2 at the time of starting study treatment
  7. Leptomeningeal metastases
  8. Spinal cord compression or brain metastases unless asymptomatic, treated and stable, and not requiring steroids within 4 weeks prior to study treatment initiation
  9. Clinically significant abnormalities of glucose metabolism as defined by any of the following:

     a. HbA1c ≥8.0% (63.9 mmol/mol) at screening. Note: for any patient with evidence of impaired glucose control or insulin resistance refer to the Capivasertib Toxicity Management Guidelines.
  10. Inadequate bone marrow reserve or organ function as demonstrated by any of the following laboratory values:

      1. Absolute neutrophil count <1.5 × 109/L
      2. Platelet count <100 × 109/L
      3. Haemoglobin <9 g/dL (<5.59 mmol/L). [NOTE: any blood transfusion must be >14 days prior to the determination of a haemoglobin ≥9 g/dL (≥5.59 mmol/L)]
      4. Alanine aminotransferase (ALT) and Aspartate aminotransferase (AST) >2.5 times upper limit of normal (ULN) if no demonstrable liver metastases or >5 × ULN in the presence of liver metastases
      5. Total bilirubin >1.5 × ULN (Patients with confirmed Gilbert's syndrome may be included in the study)
      6. Creatinine >1.5 × ULN concurrent with creatinine clearance <50 mL/min (measured or calculated by Cockcroft and Gault equation); creatinine clearance is only required when creatinine is >1.5 × ULN
  11. Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension, or active infection including tuberculosis, hepatitis B, hepatitis C, and human immunodeficiency virus (HIV), including those who have confirmed COVID 19 and any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that, in the investigator's opinion, gives reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug, may affect the interpretation of the results, render the patient at high risk from treatment complications or interferes with obtaining informed consent. Screening for chronic conditions is not required.

      Note: Known active hepatitis B or C infection, positive hepatitis C antibody, positive hepatitis B virus surface antigen. Participants positive for HCV antibody are eligible only if polymerase chain reaction is negative for HCV RNA. Patients receiving antiretroviral therapies which are strong inhibitors or inducers of CYP3A4 will be excluded due to the potential for drug-drug interaction with capivasertib
  12. Known abnormalities in coagulation such as bleeding diathesis, or treatment with anticoagulants precluding intramuscular injections of fulvestrant or subcutaneous injections of GNRH agonist (if applicable)
  13. Refractory nausea and vomiting, malabsorption syndrome, chronic gastrointestinal diseases, inability to swallow the formulated product or previous significant bowel resection, or other condition that would preclude adequate absorption of capivasertib
  14. Previous allogenic bone marrow or solid organ transplant
  15. History of another primary malignancy
  16. Known immunodeficiency syndrome
  17. Mean resting corrected QT interval >470 ms, obtained from triplicate ECGs performed at screening. History of QT prolongation associated with other medications that required discontinuation of that medication [Congenital long QT syndrome, family history of long QT syndrome, or unexplained sudden death under 40 years of age in first-degree relatives.]
  18. Medical history significant for arrhythmia (e.g., multifocal premature ventricular contractions, bigeminy, trigeminy, ventricular tachycardia), which is symptomatic or requires treatment (CTCAE Grade 3), symptomatic or uncontrolled atrial fibrillation despite treatment, or asymptomatic sustained ventricular tachycardia. Participants with atrial fibrillation controlled by medication or arrhythmias controlled by pacemakers may be permitted to enter the study based on the Investigator judgement with cardiologist consultation recommended.
  19. Any factors that increase the risk of QTc prolongation or risk of arrhythmic events, hypokalaemia of Grade >1, potential for Torsades de Pointes, congenital long QT syndrome
  20. Experience of any of the following procedures or conditions in the preceding 3 months: coronary artery bypass graft, angioplasty, myocardial infarction, unstable angina pectoris. Congestive heart failure New York Heart Association (NYHA) ≥grade 2.
  21. History of hypersensitivity to active or inactive excipients of capivasertib, fulvestrant and GNRH agonists (if applicable, i.e., concomitant GNRH agonist required in this study) or drugs with a similar chemical structure or class to capivasertib, fulvestrant or GNRH agonists (if applicable)
  22. Radiotherapy within 14 days prior to first dose of capivasertib
  23. Major surgical procedure (excluding placement of vascular access) or significant traumatic injury within 4 weeks of the first dose of study intervention or an anticipated need for major surgery during the study.
  24. Evidence of dementia altered mental status or any psychiatric condition that would prohibit understanding or rendering of informed consent
  25. Pregnancy or breastfeeding
  26. Patients who at time of data collection for this study are participating in or have participated in an interventional study that remains blinded
  27. More than 2 lines of endocrine-based therapy for inoperable locally advanced or mBC
  28. More than 1 line of chemotherapy for inoperable locally advanced or mBC. Adjuvant and neoadjuvant chemotherapy are not classed as lines of chemotherapy for mBC
  29. Prior treatment with any of the following:

      1. AKT, PIK3 and mTOR inhibitors
      2. ngSERD (Note: prior treatment with fulvestrant (=SERD) is allowed!)
      3. Nitrosourea or mitomycin C within 6 weeks prior to study treatment initiation
      4. Any other chemotherapy, immunotherapy, immunosuppressant medication (other than corticosteroids) or anticancer agents within 3 weeks prior to study treatment initiation. A longer washout period may be required for drugs with a long half-life (e.g., biologics) as agreed by the sponsor
      5. Potent inhibitors or inducers of CYP3A4 within 2 weeks prior to the first dose of study treatment (3 weeks for St John's wort) or drugs that are sensitive to CYP3A4 inhibition within 1 week prior to study treatment initiation.
      6. Any concomitant medication that may interfere with capivasertib or fulvestrant safety and efficacy based on the Investigator´s Brochure of capivasertib and the prescribing information of fulvestrant and local clinical guidelines, e.g., that are known to be associated with Torsade de Pointes or potent inducers of cytochrome P450 3A4 (CYP3A4).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-11-27 (Actual); Primary Completion 2030-03 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
Superiority* of TTNT1 in patients receiving capivasertib compared to an evidence-based "standard TTNT1 curve" for patients without capivasertib. | Last-patient-in plus 12 months
  * Statistical comparison by survival modelling of time on treatment including competing risks.
  * Standard curve is derived from placebo + fulvestrant arm of CAPItello-291 trial and corresponds to 17% remaining "on-treatment" at 12 months.
  * Stratification by eHealth support vs. no eHealth support
Superiority* of PRO-adherence compared to non-adherence regarding TTDQoL (aka DQoL-free interval). | through study completion, after 170 total DQoL-events occurred
  * The event DQoL is defined in terms of a 10-point drop of the FACT-G score compared to baseline.
  * A patient is classified here as "PRO-non-adherent" if she does not use CANKADO on 60 or more of the first 90 days, otherwise as "PRO-adherent".

SECONDARY OUTCOMES:
Progression-free survival (PFS): defined by either: • evidence of disease progression as assessed by treating physician or • death | From date of inclusion until the date of first documented progression, assessed up to 60 months
  • To evaluate progression-free survival (PFS) from index date (CAPI initiation)
Overall survival (OS) | From date of inclusion until the date of first documented progression, assessed up to 60 months
  • To evaluate overall survival (OS) from index date
Superiority of eHealth support (and summary statistics) regarding TTDQoL compared to patients entering the trial without eHealth support.** | From date of inclusion until the date of first documented progression, assessed up to 60 months
  • To evaluate the impact of eHealth support (with or without PRO-adherence) compared to no eHealth support regarding the DQoL-free interval (TTDQoL as defined above)
Evaluation of prophylactic and reactive treatments for AESI management | Treatment start until end of study, assessed up to 60 months
  • To characterise the management of AESIs

OTHER OUTCOMES:
Adverse Events with Common Terminology Criteria for Adverse Events (CTCAE) version 5 grade 3 and 4 | Treatment start until end of study, assessed up to 60 months
  • AE with CTCAE v5 grade 3+4
Adverse Events of Specila Interest (AESI)-rate | Treatment start until end of study, assessed up to 60 months
  • AESI-rate

CONTACTS AND LOCATIONS:
Overall Officials: Peter Schmid, PHD Dr, Principal Investigator — Westdeutsche Studiengruppe GmbH
Locations (7):
- Belgium (2):
  - Institut Jules Bordet, Anderlecht
  - CHC MontLegia, Liège
- Germany (4):
  - St. Elisabeth-Krankenhaus GmbH, Brustzentrum - Senologie, Cologne, North Rhine-Westphalia
  - Universitätsklinikum Essen, Essen, North Rhine-Westphalia
  - Brustzentrum Niederrhein, Johanniter Bethesda Krankenhaus, Mönchengladbach, North Rhine-Westphalia
  - Universitätsklinikum Münster AöR Brustzentrum, Münster, North Rhine-Westphalia
- Champalimaud Clinical Centre, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No